CLINICAL TRIAL: NCT03884777
Title: Incidence and Risk of Influenza in Myasthenic Patients Hospitalized in Intensive Care
Brief Title: Incidence and Risk of Influenza in Myasthenic Patients
Status: Completed | Type: Observational
Sponsor: Centre d'Investigation Clinique et Technologique 805 (Other)
Responsible Party: Sponsor
Other Study IDs: CIC1429
Record Dates: First submitted 2019-01-16; First posted 2019-03-21 (Actual); Last update posted 2019-03-21 (Actual); Status verified 2017-12

CONDITIONS: Myasthenic Crisis; Upper Respiratory Infection
Keywords: Influenza A virus; myasthenia gravis; neurocritical care clinical; neuromuscular disease
MeSH Terms: conditions — Respiratory Tract Infections; Myasthenia Gravis; Neuromuscular Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Upper respiratory infection , including influenza, may exacerbate the symptoms of myasthenia gravis (MG), which is an autoimmune disease that causes muscle weakness and, in some cases, can precipitate a myasthenic crisis

In the present study, we investigated the incidence and risk factors of influenza infection on in myasthenia gravis patients.

DETAILED DESCRIPTION:
This is a descriptive study. The data will be analyzed retrospectively . Inclusion of 416 cases of influenza in myasthenic patients treated in the intensive care unit of Garches Hospital between January 1, 2009 and December 31, 2017.

Patients who meet the inclusion and non inclusion criteria and do not object to participate in the study will be collected in a database for analysis.

ELIGIBILITY:
Inclusion Criteria:

* Men or women over the age of 18.
* Myasthenic patients hospitalized in intensive care.
* Patients with confirmed influenza infection

Exclusion Criteria:

* Age <18 years,
* Other neuromuscular diseases,
* Patient opposing the use of his data

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Inclusion of 416 cases of myasthenic patients treated in the intensive care unit of Garches Hospital between January 1, 2009 and December 31, 2017.
Sampling Method: Non-Probability Sample
Enrollment: 400 (Actual)
Dates: Start 2009-01-01 (Actual); Primary Completion 2017-12-31 (Actual); Study Completion 2017-12-31 (Actual)

PRIMARY OUTCOMES:
Incidence of influenza in myasthenic patient in crisis | between January 1, 2009 and December 31, 2017.
  Number of influenza cases in myasthenic patients

SECONDARY OUTCOMES:
Risk factors for poor outcomes | between January 1, 2009 and December 31, 2017.
  To identify risk factors for severe influenza in myasthenic patients

CONTACTS AND LOCATIONS:
Overall Officials: Rania BOUNAB, Dr, Study Director — Raymond Poincaré Hospital

REFERENCES:
- [Result] Petrova VN, Russell CA. The evolution of seasonal influenza viruses. Nat Rev Microbiol. 2018 Jan;16(1):60. doi: 10.1038/nrmicro.2017.146. Epub 2017 Nov 7. PMID 29109554
- [Result] Tackenberg B, Schneider M, Blaes F, Eienbroker C, Schade-Brittinger C, Wellek A, Deschauer M, Eickmann M, Klenk HD, Muller HH, Sommer N. Acetylcholine Receptor Antibody Titers and Clinical Course after Influenza Vaccination in Patients with Myasthenia Gravis: A Double-Blind Randomized Controlled Trial (ProPATIent-Trial). EBioMedicine. 2018 Feb;28:143-150. doi: 10.1016/j.ebiom.2018.01.007. Epub 2018 Jan 10. PMID 29337134
- [Result] Friman G, Schiller HH, Schwartz M. Distubed neuromuscular transmission in viral infections. Scand J Infect Dis. 1977;9(2):99-103. doi: 10.3109/inf.1977.9.issue-2.08. PMID 197596
- [Result] Rosciszewska D, Bluszcz M, Kurek H. [Antibodies for DNA and RNA viruses in the serum of myasthenia patients. Preliminary report]. Neurol Neurochir Pol. 1981 Sep-Dec;15(5-6):541-4. Polish. PMID 6281675